CLINICAL TRIAL: NCT00148850
Title: A Randomized, Phase 3, Double Blind, Multicentre Trial, Evaluating the Effect of Pioglitazone Versus Placebo on Change in Lipoatrophy in HIV- 1 Infected Patients Treated With Stable Antiretroviral Therapy for at Least 6 Months.ANRS 113 LIPIOT Study
Brief Title: Effect of Pioglitazone on HIV-1 Related Lipoatrophy: a Randomized, Double Blind, Placebo-Controlled Trial in 130 Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANRS 113 LIPIOT
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2005-09

CONDITIONS: HIV-Associated Lipodystrophy Syndrome; HIV Infections
Keywords: HIV-Associated Lipodystrophy Syndrome; pioglitazone; HIV infections; Treatment Experienced
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; HIV Infections | interventions — Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
The aim of this randomized study is to compare the effect of pioglitazone versus placebo on change in limb fat in HIV 1-infected patients treated with antiretroviral therapy for at least 6 months and with clinical lipoatrophy.

DETAILED DESCRIPTION:
Lipodystrophy is one of the most frequent treatment side effect in HIV-1 infected patients. This complication can be stigmatizing in some affected patients and lead to reduced adherence to treatment, increased risk of cardiovascular complications and induce insulinoresistance. The pathophysiology of lipodystrophy remains poorly understood. Some antiretroviral drugs could be involved. Therefore, using PPAR G as a therapeutic target with the objective to reverse drug induced lipoatrophy appeared as a promising objective Thiazolidinediones are a new class of insulin sensitizing drugs for the treatment of type 2 diabetes. These PPARG agonist which mainly promote the differentiation of adipocytes, decrease circulating plasma free fatty acids. In non-HIV infected patients this class of drugs decreases intraabdominal fat accumulation and increases subcutaneous fat depot.

Different previous studies were performed with that aim, most of them using rosiglitazone.

We designed a prospective randomized, double blind placebo controlled multicentre study aiming to test the hypothesis that pioglitazone would improve lipoatrophy without deleterious effect on lipid profile in adult subjects receiving antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of ages and older
* Confirmed laboratory diagnosis of HIV-1-infection
* Karnofsky equal or over 70%
* Patients treated with stable antiretroviral therapy for at least 6 months
* Plasma viral load below 400 copies/ ml and CD4 count over 200/mm3 for at least 6 months
* Patients with a clinical peripheral lipoatrophy self reported by the patient and confirmed by physical examination

Exclusion Criteria:

* Cachexia
* Cardiac failure class3 or 4 at NYHA classification
* Acute opportunistic infection
* Pregnancy or breast-feeding
* Polynuclear neutrophils below 1000/mm3
* Hemoglobin below 9 g/dl
* Platelets below 50 000/mm3
* Creatinine level over 2 UN
* ASAT, ALAT over 2.5UN
* Bilirubin, amylase, lipase level over 2 UN
* CD4 count below 200/mm3
* Patients treated by any antidiabetic or lipid lowering drugs, anabolic or corticosteroid hormone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-02; Study Completion 2004-10

PRIMARY OUTCOMES:
Evolution from inclusion to week 48 of limb fat using DEXA Scan (Dual Energy X-ray Absorptiometry)

SECONDARY OUTCOMES:
Changes from inclusion to week 48:
Lipid profile and the glucidic metabolism
SAT/TAT and VAT/TAT ratios evaluated with scanner
X ray of L4
Anthropometric measurements and the quality of life (WHO-QOL-HIV BREF)
Evaluation of clinical and biological safety

CONTACTS AND LOCATIONS:
Overall Officials: Willy Rozenbaum, MD, Principal Investigator — Hopital Tenon Paris; Dominique Costagliola, Study Chair — INSERM U 720
Locations (1):
- Service des Maladies Infectieuses et Tropicales, Hopital Tenon, Paris, France

REFERENCES:
- [Derived] Slama L, Lanoy E, Valantin MA, Bastard JP, Chermak A, Boutekatjirt A, William-Faltaos D, Billaud E, Molina JM, Capeau J, Costagliola D, Rozenbaum W. Effect of pioglitazone on HIV-1-related lipodystrophy: a randomized double-blind placebo-controlled trial (ANRS 113). Antivir Ther. 2008;13(1):67-76. PMID 18389900